CLINICAL TRIAL: NCT05556148
Title: A Real-World Evidence Study Evaluating Quality of Life Parameters Following Treatment With Otrivine (Xylometazoline Hydrochloride)
Brief Title: Otrivine: Quality of Life (QoL) Impact in a Real-World Setting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 218317
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Results first posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Common Cold
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Otrivine Congestion Relief (Experimental): Participants will be instructed to use the product per label and leaflet instructions: 1 spray in each nostril up to 3 times per day until resolution of symptoms or up to a maximum of 7 days, whichever occurs first.
  Interventions: Drug: Otrivine Congestion Relief

INTERVENTIONS:
Drug: Otrivine Congestion Relief — 0.1% Nasal Spray (Xylometazoline Hydrochloride)

SUMMARY:
This study is designed to generate real world data from participants with nasal congestion acquired from common cold following treatment with a marketed nasal spray. The main purpose of this study is to evaluate the effectiveness of a nasal spray on quality of life (QoL) factors.

DETAILED DESCRIPTION:
This is a longitudinal, open-label study evaluating the effect on QoL factors in participants with the common cold using Otrivine nasal spray (xylometazoline hydrochloride 0.1 percent [%]), in a real-world setting. A sufficient number of adults aged 18 years and over with symptoms of common cold will be screened for eligibility. The study expects to enroll approximately 125 participants to ensure that 100 participants complete the study. All study data will be collected remotely through a study app using the participant's own mobile device.

ELIGIBILITY:
Inclusion Criteria:

* Participant's provision of a signed and dated electronic informed consent (eIC) form indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Participant reporting a nasal congestion, and at least another common cold symptom among runny nose, sore throat, cough.
* Participant reporting a minimum score of 5 (moderate) for plugged nose associated with common cold symptoms and at least one other symptom of common cold (at least mild score of 3) as per the WURSS-21 questionnaire at screening.
* Participant reporting initiation of cold symptoms within no longer than 24 hours of prior to initiation of screening.
* Participants confirm common cold symptoms within 24 hours of study product receipt of minimum score of 5 (moderate) for plugged nose associated with common cold symptoms and at least one other symptom of common cold (at least mild score of 3) as per the WURSS-21 questionnaire.
* Male and female Participants.
* Participant that owns a smart device and willing to download the study app.
* Participant who is willing and able to complete all activities as shown in the Schedule of Activities independently on own smart devices.
* Participant is in good general and mental health.
* Participant who has a self-reported medical diagnosis of cardiovascular disease (including those with long QT syndrome), hyperthyroidism or diabetes mellitus, may be included if deemed acceptable by a medically qualified investigator.
* Participant who is showing a strong reaction to adrenergic substances, as manifested by signs of insomnia, dizziness, tremor, cardiac arrhythmias, or elevated blood pressure, may be included if deemed acceptable by a medically qualified investigator.

Exclusion Criteria:

* Participants under 18 years of age.
* Participants who are allergic to xylometazoline hydrochloride or any of the other ingredients in the spray (see product label).
* Participants who have had recent neurosurgery.
* Participants who self-report narrow angle glaucoma, chronic nasal inflammation with very dry nasal passages (rhinitis sicca or atrophic rhinitis), or enlarged prostate gland.
* Participants who self-report a rare tumor of the adrenal gland that produces high amounts of adrenaline and noradrenaline (phaeochromocytoma).
* Participants who are taking monoamine oxidase inhibitors (MAOIs) or have stopped taking them in the last 14 days.
* Participants who are pregnant, lactating, or plan to be pregnant or lactating during the course of the study.
* Participant who is currently using or has used a nasal decongestant (for example, adrenergic, steroids) within the last 7 days (or for more than 7 days) prior to initiating study treatment.
* Participants who have tested positive for COVID-19 within one month prior to enrollment into the study.
* Participants who have taken a vaccine one week prior to enrollment into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The VCTC, Swadlincote, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.

REFERENCES:
- [Derived] Hagen M, Clark K, Kalita P, Serra G, Sanchez E, Varbiro G, Albasser MM. A real-world study of quality of life following treatment with xylometazoline hydrochloride in individuals with common cold. Ther Adv Respir Dis. 2024 Jan-Dec;18:17534666241228927. doi: 10.1177/17534666241228927. PMID 38372128

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a decentralized study in participants with common cold using Otrivine nasal spray (xylometazoline hydrochloride 0.1 percent [%]), in a real-world setting. Participants were recruited through targeted advertising on social media channels. All study data were collected remotely through a study app using the participant's own mobile device.
Pre-assignment Details: A total of 172 participants were screened of which 136 were enrolled and 100 completed the study. A total of 36 participants were discontinued from the study.
Groups:
- Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride): Participants were instructed to use Otrivine congestion relief 0.1% nasal spray (xylometazoline hydrochloride) per label and leaflet instructions. Participants administered 1 spray in each nostril up to 3 times per day until resolution of symptoms or up to a maximum of 7 days, whichever occurred first.
Period: Overall Study
Arm/Group | Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride)
Started | 136
Modified Intent-To-Treat (mITT) Population (The mITT population included all participants who used study product at least once and had data from at least one post-baseline quality of life (QoL) questionnaire to support at least one of the primary endpoint assessments.) | 102
Completed | 100
Not Completed | 36
Not completed — Early Termination | 29
Not completed — Baseline Tasks Expired | 4
Not completed — Family Emergency: Could no longer take part | 1
Not completed — No Longer Wished to Participate | 1
Not completed — Bacterial Conjunctivitis | 1

BASELINE CHARACTERISTICS:
Population: The mITT population included all participants who used study product at least once and had data from at least one post-baseline QoL questionnaire to support at least one of the primary endpoint assessments.
Arm/Group | Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride)
Number analyzed (Participants) | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (12.04)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 73
  Male | 25
  Other | 2
  Prefer not to tell | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 99
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian or Asian British | 18
  Black, Black British, Caribbean or African | 1
  White | 78
  Mixed or Multiple Ethnic Groups | 3
  Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Wisconsin Upper Respiratory Symptom Survey-21 (WURSS-21) Total Score
Description: The WURSS is an evaluative illness specific quality of life instrument, designed to assess the negative impact of acute upper respiratory infection, presumed viral (the common cold). WURSS-21 is the short version of this validated survey. Participants rated their cold symptoms and QoL related questions using WURSS-21. It consisted of 10 symptoms questions and 9 QoL questions, the responses of which were evaluated on a scale ranging from 0 to 7, where 0=Do not have symptoms/Not at all and 7=Severe symptoms/Severely. Thus, the minimum and maximum possible total scores were 0 and 133 respectively, where higher total scores indicated more negative impact on symptoms and quality of life. Baseline was defined as Day 0. Change from Baseline was calculated as each post-Baseline value minus Baseline value. A negative change from Baseline indicated improvement in symptoms and quality of life.
Time Frame: Baseline (Day 0) up to Day 7
Population: The mITT population included all participants who used study product at least once and had data from at least one post-baseline QoL questionnaire to support at least one of the primary endpoint assessments. Only those participants with data available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride): Participants were instructed to use Otrivine congestion relief 0.1% nasal spray (xylometazoline hydrochloride) per label and leaflet instructions. Participants administered 1 spray in each nostril up to 3 times per day until resolution of symptoms or up to a maximum of 7 days, whichever occured first.
Arm/Group | Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride)
Number analyzed (Participants) | 102
score on a scale
  Baseline | 75.8 (20.23)
  Change from Baseline at Day 1: number analyzed (Participants) | 99
  Change from Baseline at Day 1 | -1.5 (14.57)
  Change from Baseline at Day 2: number analyzed (Participants) | 98
  Change from Baseline at Day 2 | -15.4 (22)
  Change from Baseline at Day 3: number analyzed (Participants) | 92
  Change from Baseline at Day 3 | -27.3 (27.94)
  Change from Baseline at Day 4: number analyzed (Participants) | 82
  Change from Baseline at Day 4 | -35.0 (30.21)
  Change from Baseline at Day 5: number analyzed (Participants) | 59
  Change from Baseline at Day 5 | -38.5 (28.31)
  Change from Baseline at Day 6: number analyzed (Participants) | 39
  Change from Baseline at Day 6 | -39.7 (27.12)
  Change from Baseline at Day 7: number analyzed (Participants) | 30
  Change from Baseline at Day 7 | -52.6 (29.7)
Statistical Analysis 1: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 1; Test type: Other; p = 0.2968, Student's paired t-test; Mean Difference (Final Values) = -1.54, 95% CI 2-sided [-4.44 to 1.37]
Statistical Analysis 2: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 2; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -15.36, 95% CI 2-sided [-19.77 to -10.95]
Statistical Analysis 3: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 3; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -27.27, 95% CI 2-sided [-33.06 to -21.49]
Statistical Analysis 4: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 4; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -35.05, 95% CI 2-sided [-41.69 to -28.41]
Statistical Analysis 5: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 5; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -38.49, 95% CI 2-sided [-45.87 to -31.11]
Statistical Analysis 6: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 6; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -39.67, 95% CI 2-sided [-48.46 to -30.88]
Statistical Analysis 7: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 7; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -52.60, 95% CI 2-sided [-63.69 to -41.51]

2. Primary Outcome: Change From Baseline in WURSS-21 Total Symptom Domains Score
Description: The WURSS is an evaluative illness specific quality of life instrument, designed to assess the negative impact of acute upper respiratory infection, presumed viral (the common cold). WURSS-21 is the short version of this validated survey. The symptom domain of WURSS-21 consisted of 10 questions. Participants rated their cold symptoms related questions, the responses of which were evaluated on a scale ranging from 0 to 7, where 0=Do not have symptoms and 7=Severely. Thus, the minimum and maximum possible total score were 0 and 70 respectively, where higher scores indicated a negative impact on symptoms. Baseline was defined as Day 0. Change from Baseline was calculated as each post-Baseline value minus Baseline value. A negative change from Baseline indicated improvement of symptoms.
Time Frame: Baseline (Day 0) up to Day 7
Population: mITT population. Only those participants with data available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride)
Number analyzed (Participants) | 102
score on a scale
  Baseline | 38.3 (11.35)
  Change from Baseline at Day 1: number analyzed (Participants) | 99
  Change from Baseline at Day 1 | 0.3 (7.85)
  Change from Baseline at Day 2: number analyzed (Participants) | 98
  Change from Baseline at Day 2 | -6.2 (11.44)
  Change from Baseline at Day 3: number analyzed (Participants) | 92
  Change from Baseline at Day 3 | -12.1 (13.96)
  Change from Baseline at Day 4: number analyzed (Participants) | 82
  Change from Baseline at Day 4 | -16.0 (14.88)
  Change from Baseline at Day 5: number analyzed (Participants) | 59
  Change from Baseline at Day 5 | -19.4 (14.77)
  Change from Baseline at Day 6: number analyzed (Participants) | 39
  Change from Baseline at Day 6 | -19.4 (14.4)
  Change from Baseline at Day 7: number analyzed (Participants) | 30
  Change from Baseline at Day 7 | -25.4 (17.32)
Statistical Analysis 1: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 1; Test type: Other; p = 0.7112, Student's paired t-test; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [-1.27 to 1.86]
Statistical Analysis 2: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 2; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -6.21, 95% CI 2-sided [-8.51 to -3.92]
Statistical Analysis 3: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 3; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -12.11, 95% CI 2-sided [-15.00 to -9.22]
Statistical Analysis 4: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 4; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -15.98, 95% CI 2-sided [-19.24 to -12.71]
Statistical Analysis 5: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 5; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -19.44, 95% CI 2-sided [-23.29 to -15.59]
Statistical Analysis 6: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 6; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -19.36, 95% CI 2-sided [-24.03 to -14.69]
Statistical Analysis 7: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 7; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -25.40, 95% CI 2-sided [-31.87 to -18.93]

3. Primary Outcome: Change From Baseline in WURSS-21 Total QoL Domains Score
Description: The WURSS is an evaluative illness specific quality of life instrument, designed to assess the negative impact of acute upper respiratory infection, presumed viral (the common cold). WURSS-21 is the short version of this validated survey. The QoL domain of WURSS-21 consisted of 9 questions. Participants rated their QoL related questions, the responses of which were evaluated on a scale ranging from 0 to 7, where 0=Not at all and 7=Severely. Thus, the minimum and maximum possible total scores were 0 and 63 respectively, where higher scores indicated a negative impact on QoL. Baseline was defined as Day 0. Change from Baseline was calculated as each post-Baseline value minus Baseline value. A negative change from Baseline indicated improvement of quality of life.
Time Frame: Baseline (Day 0) up to Day 7
Population: mITT population. Only those participants with data available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride)
Number analyzed (Participants) | 102
score on a scale
  Baseline | 37.5 (11.61)
  Change From Baseline at Day 1: number analyzed (Participants) | 99
  Change From Baseline at Day 1 | -1.8 (9.09)
  Change From Baseline at Day 2: number analyzed (Participants) | 98
  Change From Baseline at Day 2 | -9.1 (12.95)
  Change From Baseline at Day 3: number analyzed (Participants) | 92
  Change From Baseline at Day 3 | -15.2 (15.84)
  Change From Baseline at Day 4: number analyzed (Participants) | 82
  Change From Baseline at Day 4 | -19.1 (17.17)
  Change From Baseline at Day 5: number analyzed (Participants) | 59
  Change From Baseline at Day 5 | -19.1 (16.5)
  Change From Baseline at Day 6: number analyzed (Participants) | 39
  Change From Baseline at Day 6 | -20.3 (16.62)
  Change From Baseline at Day 7: number analyzed (Participants) | 30
  Change From Baseline at Day 7 | -27.2 (14.14)
Statistical Analysis 1: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 1; Test type: Other; p = 0.0481, Student's paired t-test; Mean Difference (Final Values) = -1.83, 95% CI 2-sided [-3.64 to -0.02]
Statistical Analysis 2: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 2; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -9.14, 95% CI 2-sided [-11.74 to -6.55]
Statistical Analysis 3: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 3; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -15.16, 95% CI 2-sided [-18.44 to -11.88]
Statistical Analysis 4: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 4; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -19.07, 95% CI 2-sided [-22.84 to -15.30]
Statistical Analysis 5: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 5; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -19.05, 95% CI 2-sided [-23.35 to -14.75]
Statistical Analysis 6: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 6; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -20.31, 95% CI 2-sided [-25.70 to -14.92]
Statistical Analysis 7: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 7; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -27.20, 95% CI 2-sided [-32.48 to -21.92]

4. Primary Outcome: Change From Baseline in Each of the WURSS-21 Symptom Domains Score: Runny Nose
Description: The WURSS is an evaluative illness specific quality of life instrument, designed to assess the negative impact of acute upper respiratory infection, presumed viral (the common cold). WURSS-21 is the short version of this validated survey. The individual symptoms included runny nose, plugged nose, sneezing, sore throat, scratchy throat, cough, hoarseness, head congestion, chest congestion and feeling tired. Participants rated each of the 10 individual symptom domain questions, the responses of which were evaluated on a scale ranging from 0 to 7, where 0=Do not have symptom and 7=Severely. Thus, the minimum and maximum score for each symptom domain question were 0 and 7, where higher scores indicated a negative impact on symptoms. Baseline was defined as Day 0. Change from Baseline was calculated as each post-Baseline value minus Baseline value. A negative change from Baseline indicated improvement in symptom.
Time Frame: Baseline (Day 0) up to Day 7
Population: mITT population. Only those participants with data available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride)
Number analyzed (Participants) | 102
score on a scale
  Baseline | 4.0 (1.86)
  Change from Baseline at Day 1: number analyzed (Participants) | 99
  Change from Baseline at Day 1 | 0.0 (1.53)
  Change from Baseline at Day 2: number analyzed (Participants) | 98
  Change from Baseline at Day 2 | -0.6 (1.68)
  Change from Baseline at Day 3: number analyzed (Participants) | 92
  Change from Baseline at Day 3 | -1.1 (1.93)
  Change from Baseline at Day 4: number analyzed (Participants) | 82
  Change from Baseline at Day 4 | -1.7 (2.20)
  Change from Baseline at Day 5: number analyzed (Participants) | 59
  Change from Baseline at Day 5 | -1.7 (2.24)
  Change from Baseline at Day 6: number analyzed (Participants) | 39
  Change from Baseline at Day 6 | -1.9 (1.90)
  Change from Baseline at Day 7: number analyzed (Participants) | 30
  Change from Baseline at Day 7 | -2.5 (2.21)
Statistical Analysis 1: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 1; Test type: Other; p = 1.0000, Student's paired t-test; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.31 to 0.31]
Statistical Analysis 2: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 2; Test type: Other; p = 0.0003, Student's paired t-test; Mean Difference (Final Values) = -0.63, 95% CI 2-sided [-0.97 to -0.30]
Statistical Analysis 3: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 3; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -1.10, 95% CI 2-sided [-1.50 to -0.70]
Statistical Analysis 4: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 4; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -1.72, 95% CI 2-sided [-2.20 to -1.24]
Statistical Analysis 5: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 5; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -1.75, 95% CI 2-sided [-2.33 to -1.16]
Statistical Analysis 6: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 6; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -1.90, 95% CI 2-sided [-2.51 to -1.28]
Statistical Analysis 7: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 7; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.47, 95% CI 2-sided [-3.29 to -1.64]

5. Primary Outcome: Change From Baseline in Each of the WURSS-21 Symptom Domains Score: Plugged Nose
Description: as for outcome 4
Time Frame: Baseline (Day 0) up to Day 7
Population: mITT population. Only those participants with data available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride)
Number analyzed (Participants) | 102
score on a scale
  Baseline | 5.5 (0.92)
  Change From Baseline at Day 1: number analyzed (Participants) | 99
  Change From Baseline at Day 1 | -0.4 (1.25)
  Change From Baseline at Day 2: number analyzed (Participants) | 98
  Change From Baseline at Day 2 | -1.5 (1.75)
  Change From Baseline at Day 3: number analyzed (Participants) | 92
  Change From Baseline at Day 3 | -2.0 (1.99)
  Change From Baseline at Day 4: number analyzed (Participants) | 82
  Change From Baseline at Day 4 | -2.4 (1.95)
  Change From Baseline at Day 5: number analyzed (Participants) | 59
  Change From Baseline at Day 5 | -3.0 (1.94)
  Change From Baseline at Day 6: number analyzed (Participants) | 39
  Change From Baseline at Day 6 | -2.8 (1.83)
  Change From Baseline at Day 7: number analyzed (Participants) | 30
  Change From Baseline at Day 7 | -3.3 (2.06)
Statistical Analysis 1: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 1; Test type: Other; p = 0.0023, Student's paired t-test; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-0.64 to -0.14]
Statistical Analysis 2: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 2; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -1.47, 95% CI 2-sided [-1.82 to -1.12]
Statistical Analysis 3: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 3; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -1.99, 95% CI 2-sided [-2.40 to -1.58]
Statistical Analysis 4: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 4; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.43, 95% CI 2-sided [-2.86 to -2.00]
Statistical Analysis 5: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 5; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -3.00, 95% CI 2-sided [-3.51 to -2.49]
Statistical Analysis 6: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 6; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.77, 95% CI 2-sided [-3.36 to -2.18]
Statistical Analysis 7: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 7; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -3.33, 95% CI 2-sided [-4.10 to -2.57]

6. Primary Outcome: Change From Baseline in Each of the WURSS-21 Symptom Domains Score: Sneezing
Description: as for outcome 4
Time Frame: Baseline (Day 0) up to Day 7
Population: mITT population. Only those participants with data available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride)
Number analyzed (Participants) | 102
score on a scale
  Baseline | 3.6 (1.80)
  Change From Baseline at Day 1: number analyzed (Participants) | 99
  Change From Baseline at Day 1 | -0.1 (1.46)
  Change From Baseline at Day 2: number analyzed (Participants) | 98
  Change From Baseline at Day 2 | -0.9 (1.62)
  Change From Baseline at Day 3: number analyzed (Participants) | 92
  Change From Baseline at Day 3 | -1.2 (1.86)
  Change From Baseline at Day 4: number analyzed (Participants) | 82
  Change From Baseline at Day 4 | -1.6 (2.14)
  Change From Baseline at Day 5: number analyzed (Participants) | 59
  Change From Baseline at Day 5 | -1.9 (2.05)
  Change From Baseline at Day 6: number analyzed (Participants) | 39
  Change From Baseline at Day 6 | -1.8 (1.87)
  Change From Baseline at Day 7: number analyzed (Participants) | 30
  Change From Baseline at Day 7 | -2.5 (1.93)
Statistical Analysis 1: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 1; Test type: Other; p = 0.4495, Student's paired t-test; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.40 to 0.18]
Statistical Analysis 2: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 2; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -0.87, 95% CI 2-sided [-1.19 to -0.54]
Statistical Analysis 3: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 3; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -1.21, 95% CI 2-sided [-1.59 to -0.82]
Statistical Analysis 4: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 4; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -1.59, 95% CI 2-sided [-2.05 to -1.12]
Statistical Analysis 5: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 5; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -1.86, 95% CI 2-sided [-2.40 to -1.33]
Statistical Analysis 6: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 6; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -1.85, 95% CI 2-sided [-2.45 to -1.24]
Statistical Analysis 7: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 7; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.47, 95% CI 2-sided [-3.19 to -1.75]

7. Primary Outcome: Change From Baseline in Each of the WURSS-21 Symptom Domains Score: Sore Throat
Description: The WURSS is an evaluative illness specific quality of life instrument, designed to assess the negative impact of acute upper respiratory infection, presumed viral (the common cold). WURSS-21 is the short version of this validated survey. The individual symptoms included runny nose, plugged nose, sneezing, sore throat, scratchy throat, cough, hoarseness, head congestion, chest congestion and feeling tired. Participants rated each of the 10 individual symptom domain questions, the responses of which were evaluated on a scale ranging from 0 to 7, where 0=Do not have symptom and 7=Severely. Thus, the minimum and maximum score for each symptom domain question were 0 and 7, where higher scores indicated a negative impact on each individual symptom. Baseline was defined as Day 0. Change from Baseline was calculated as each post-Baseline value minus Baseline value. A negative change from Baseline indicated improvement in symptoms.
Time Frame: Baseline (Day 0) up to Day 7
Population: mITT population. Only those participants with data available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride)
Number analyzed (Participants) | 102
score on a scale
  Baseline | 3.5 (2.05)
  Change from Baseline to Day 1: number analyzed (Participants) | 99
  Change from Baseline to Day 1 | 0.1 (1.54)
  Change from Baseline to Day 2: number analyzed (Participants) | 98
  Change from Baseline to Day 2 | -0.6 (1.86)
  Change from Baseline to Day 3: number analyzed (Participants) | 92
  Change from Baseline to Day 3 | -1.2 (2.12)
  Change from Baseline to Day 4: number analyzed (Participants) | 82
  Change from Baseline to Day 4 | -1.7 (2.33)
  Change from Baseline to Day 5: number analyzed (Participants) | 59
  Change from Baseline to Day 5 | -2.0 (1.81)
  Change from Baseline to Day 6: number analyzed (Participants) | 39
  Change from Baseline to Day 6 | -2.1 (2.13)
  Change from Baseline to Day 7: number analyzed (Participants) | 30
  Change from Baseline to Day 7 | -2.9 (2.10)
Statistical Analysis 1: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 1; Test type: Other; p = 0.4758, Student's paired t-test; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.20 to 0.42]
Statistical Analysis 2: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 2; Test type: Other; p = 0.0016, Student's paired t-test; Mean Difference (Final Values) = -0.61, 95% CI 2-sided [-0.99 to -0.24]
Statistical Analysis 3: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 3; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -1.23, 95% CI 2-sided [-1.67 to -0.79]
Statistical Analysis 4: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 4; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -1.67, 95% CI 2-sided [-2.18 to -1.16]
Statistical Analysis 5: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 5; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -1.98, 95% CI 2-sided [-2.46 to -1.51]
Statistical Analysis 6: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 6; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.08, 95% CI 2-sided [-2.77 to -1.39]
Statistical Analysis 7: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 7; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.87, 95% CI 2-sided [-3.65 to -2.08]

8. Primary Outcome: Change From Baseline in Each of the WURSS-21 Symptom Domains Score: Scratchy Throat
Description: as for outcome 4
Time Frame: Baseline (Day 0) up to Day 7
Population: mITT population. Only those participants with data available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride)
Number analyzed (Participants) | 102
score on a scale
  Baseline | 3.2 (2.11)
  Change from Baseline at Day 1: number analyzed (Participants) | 99
  Change from Baseline at Day 1 | -0.0 (1.60)
  Change from Baseline at Day 2: number analyzed (Participants) | 98
  Change from Baseline at Day 2 | -0.7 (1.86)
  Change from Baseline at Day 3: number analyzed (Participants) | 92
  Change from Baseline at Day 3 | -1.3 (1.92)
  Change from Baseline at Day 4: number analyzed (Participants) | 82
  Change from Baseline at Day 4 | -1.4 (2.04)
  Change from Baseline at Day 5: number analyzed (Participants) | 59
  Change from Baseline at Day 5 | -2.0 (1.99)
  Change from Baseline at Day 6: number analyzed (Participants) | 39
  Change from Baseline at Day 6 | -1.9 (2.03)
  Change from Baseline at Day 7: number analyzed (Participants) | 30
  Change from Baseline at Day 7 | -2.4 (2.31)
Statistical Analysis 1: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 1; Test type: Other; p = 0.8017, Student's paired t-test; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.36 to 0.28]
Statistical Analysis 2: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 2; Test type: Other; p = 0.0005, Student's paired t-test; Mean Difference (Final Values) = -0.67, 95% CI 2-sided [-1.05 to -0.30]
Statistical Analysis 3: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 3; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -1.29, 95% CI 2-sided [-1.69 to -0.89]
Statistical Analysis 4: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 4; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -1.41, 95% CI 2-sided [-1.86 to -0.97]
Statistical Analysis 5: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 5; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -1.98, 95% CI 2-sided [-2.50 to -1.47]
Statistical Analysis 6: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 6; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -1.95, 95% CI 2-sided [-2.61 to -1.29]
Statistical Analysis 7: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 7; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.40, 95% CI 2-sided [-3.26 to -1.54]

9. Primary Outcome: Change From Baseline in Each of the WURSS-21 Symptom Domains Score: Cough
Description: as for outcome 4
Time Frame: Baseline (Day 0) up to Day 7
Population: mITT population. Only those participants with data available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride)
Number analyzed (Participants) | 102
score on a scale
  Baseline | 3.3 (2.04)
  Change from Baseline at Day 1: number analyzed (Participants) | 99
  Change from Baseline at Day 1 | 0.0 (1.41)
  Change from Baseline at Day 2: number analyzed (Participants) | 98
  Change from Baseline at Day 2 | -0.4 (1.85)
  Change from Baseline at Day 3: number analyzed (Participants) | 92
  Change from Baseline at Day 3 | -0.8 (2.14)
  Change from Baseline at Day 4: number analyzed (Participants) | 82
  Change from Baseline at Day 4 | -1.0 (2.11)
  Change from Baseline at Day 5: number analyzed (Participants) | 59
  Change from Baseline at Day 5 | -1.2 (2.07)
  Change from Baseline at Day 6: number analyzed (Participants) | 39
  Change from Baseline at Day 6 | -1.1 (1.96)
  Change from Baseline at Day 7: number analyzed (Participants) | 30
  Change from Baseline at Day 7 | -1.3 (2.23)
Statistical Analysis 1: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 1; Test type: Other; p = 0.8311, Student's paired t-test; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.25 to 0.31]
Statistical Analysis 2: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 2; Test type: Other; p = 0.0313, Student's paired t-test; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-0.78 to -0.04]
Statistical Analysis 3: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 3; Test type: Other; p = 0.0003, Student's paired t-test; Mean Difference (Final Values) = -0.84, 95% CI 2-sided [-1.28 to -0.39]
Statistical Analysis 4: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 4; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -1.05, 95% CI 2-sided [-1.51 to -0.59]
Statistical Analysis 5: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 5; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -1.20, 95% CI 2-sided [-1.74 to -0.66]
Statistical Analysis 6: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 6; Test type: Other; p = 0.0018, Student's paired t-test; Mean Difference (Final Values) = -1.05, 95% CI 2-sided [-1.69 to -0.42]
Statistical Analysis 7: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 7; Test type: Other; p = 0.0041, Student's paired t-test; Mean Difference (Final Values) = -1.27, 95% CI 2-sided [-2.10 to -0.43]

10. Primary Outcome: Change From Baseline in Each of the WURSS-21 Symptom Domains Score: Hoarseness
Description: as for outcome 4
Time Frame: Baseline (Day 0) up to Day 7
Population: mITT population. Only those participants with data available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride)
Number analyzed (Participants) | 102
score on a scale
  Baseline | 2.9 (2.06)
  Change from Baseline at Day 1: number analyzed (Participants) | 99
  Change from Baseline at Day 1 | 0.0 (1.29)
  Change from Baseline at Day 2: number analyzed (Participants) | 98
  Change from Baseline at Day 2 | -0.4 (1.76)
  Change from Baseline at Day 3: number analyzed (Participants) | 92
  Change from Baseline at Day 3 | -1.0 (1.61)
  Change from Baseline at Day 4: number analyzed (Participants) | 82
  Change from Baseline at Day 4 | -1.2 (1.91)
  Change from Baseline at Day 5: number analyzed (Participants) | 59
  Change from Baseline at Day 5 | -1.8 (1.88)
  Change from Baseline at Day 6: number analyzed (Participants) | 39
  Change from Baseline at Day 6 | -1.7 (1.98)
  Change from Baseline at Day 7: number analyzed (Participants) | 30
  Change from Baseline at Day 7 | -2.3 (2.09)
Statistical Analysis 1: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 1; Test type: Other; p = 0.9380, Student's paired t-test; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.25 to 0.27]
Statistical Analysis 2: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 2; Test type: Other; p = 0.0416, Student's paired t-test; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-0.72 to -0.01]
Statistical Analysis 3: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 3; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -0.96, 95% CI 2-sided [-1.29 to -0.62]
Statistical Analysis 4: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 4; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -1.18, 95% CI 2-sided [-1.60 to -0.76]
Statistical Analysis 5: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 5; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -1.76, 95% CI 2-sided [-2.25 to -1.27]
Statistical Analysis 6: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 6; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -1.69, 95% CI 2-sided [-2.33 to -1.05]
Statistical Analysis 7: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 7; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.30, 95% CI 2-sided [-3.08 to -1.52]

11. Primary Outcome: Change From Baseline in Each of the WURSS-21 Symptom Domains Score: Head Congestion
Description: as for outcome 4
Time Frame: Baseline (Day 0) up to Day 7
Population: mITT population. Only those participants with data available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride)
Number analyzed (Participants) | 102
score on a scale
  Baseline | 4.7 (1.57)
  Change from Baseline at Day 1: number analyzed (Participants) | 99
  Change from Baseline at Day 1 | 0.0 (1.45)
  Change from Baseline at Day 2: number analyzed (Participants) | 98
  Change from Baseline at Day 2 | -0.8 (1.85)
  Change from Baseline at Day 3: number analyzed (Participants) | 92
  Change from Baseline at Day 3 | -1.6 (2.10)
  Change from Baseline at Day 4: number analyzed (Participants) | 82
  Change from Baseline at Day 4 | -2.3 (1.98)
  Change from Baseline at Day 5: number analyzed (Participants) | 59
  Change from Baseline at Day 5 | -2.5 (1.99)
  Change from Baseline at Day 6: number analyzed (Participants) | 39
  Change from Baseline at Day 6 | -2.6 (2.22)
  Change from Baseline at Day 7: number analyzed (Participants) | 30
  Change from Baseline at Day 7 | -3.2 (2.64)
Statistical Analysis 1: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 1; Test type: Other; p = 0.7821, Student's paired t-test; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.25 to 0.33]
Statistical Analysis 2: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 2; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -0.77, 95% CI 2-sided [-1.14 to -0.39]
Statistical Analysis 3: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 3; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -1.62, 95% CI 2-sided [-2.05 to -1.19]
Statistical Analysis 4: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 4; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.29, 95% CI 2-sided [-2.73 to -1.86]
Statistical Analysis 5: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 5; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.46, 95% CI 2-sided [-2.98 to -1.94]
Statistical Analysis 6: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 6; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.64, 95% CI 2-sided [-3.36 to -1.92]
Statistical Analysis 7: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 7; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -3.20, 95% CI 2-sided [-4.19 to -2.21]

12. Primary Outcome: Change From Baseline in Each of the WURSS-21 Symptom Domains Score: Chest Congestion
Description: as for outcome 4
Time Frame: Baseline (Day 0) up to Day 7
Population: mITT population. Only those participants with data available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride)
Number analyzed (Participants) | 102
score on a scale
  Baseline | 2.6 (2.07)
  Change from Baseline at Day 1: number analyzed (Participants) | 99
  Change from Baseline at Day 1 | 0.4 (1.17)
  Change from Baseline at Day 2: number analyzed (Participants) | 98
  Change from Baseline at Day 2 | -0.1 (1.53)
  Change from Baseline at Day 3: number analyzed (Participants) | 92
  Change from Baseline at Day 3 | -0.6 (1.77)
  Change from Baseline at Day 4: number analyzed (Participants) | 82
  Change from Baseline at Day 4 | -0.8 (1.90)
  Change from Baseline at Day 5: number analyzed (Participants) | 59
  Change from Baseline at Day 5 | -1.2 (1.83)
  Change from Baseline at Day 6: number analyzed (Participants) | 39
  Change from Baseline at Day 6 | -1.4 (2.11)
  Change from Baseline at Day 7: number analyzed (Participants) | 30
  Change from Baseline at Day 7 | -2.1 (2.18)
Statistical Analysis 1: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 1; Test type: Other; p = 0.0003, Student's paired t-test; Mean Difference (Final Values) = 0.44, 95% CI 2-sided [0.21 to 0.68]
Statistical Analysis 2: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 2; Test type: Other; p = 0.6460, Student's paired t-test; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.38 to 0.24]
Statistical Analysis 3: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 3; Test type: Other; p = 0.0021, Student's paired t-test; Mean Difference (Final Values) = -0.59, 95% CI 2-sided [-0.95 to -0.22]
Statistical Analysis 4: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 4; Test type: Other; p = 0.0002, Student's paired t-test; Mean Difference (Final Values) = -0.83, 95% CI 2-sided [-1.25 to -0.41]
Statistical Analysis 5: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 5; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -1.20, 95% CI 2-sided [-1.68 to -0.73]
Statistical Analysis 6: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 6; Test type: Other; p = 0.0003, Student's paired t-test; Mean Difference (Final Values) = -1.36, 95% CI 2-sided [-2.04 to -0.68]
Statistical Analysis 7: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 7; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.13, 95% CI 2-sided [-2.95 to -1.32]

13. Primary Outcome: Change From Baseline in Each of the WURSS-21 Symptom Domains Score: Feeling Tired
Description: as for outcome 4
Time Frame: Baseline (Day 0) up to Day 7
Population: mITT population. Only those participants with data available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride)
Number analyzed (Participants) | 102
score on a scale
  Baseline | 4.9 (1.60)
  Change from Baseline at Day 1: number analyzed (Participants) | 99
  Change from Baseline at Day 1 | 0.2 (1.24)
  Change from Baseline at Day 2: number analyzed (Participants) | 98
  Change from Baseline at Day 2 | -0.3 (1.62)
  Change from Baseline at Day 3: number analyzed (Participants) | 92
  Change from Baseline at Day 3 | -1.3 (1.84)
  Change from Baseline at Day 4: number analyzed (Participants) | 82
  Change from Baseline at Day 4 | -1.8 (2.05)
  Change from Baseline at Day 5: number analyzed (Participants) | 59
  Change from Baseline at Day 5 | -2.2 (2.10)
  Change from Baseline at Day 6: number analyzed (Participants) | 39
  Change from Baseline at Day 6 | -2.1 (1.92)
  Change from Baseline at Day 7: number analyzed (Participants) | 30
  Change from Baseline at Day 7 | -3.0 (2.33)
Statistical Analysis 1: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 1; Test type: Other; p = 0.1074, Student's paired t-test; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-0.04 to 0.45]
Statistical Analysis 2: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 2; Test type: Other; p = 0.0364, Student's paired t-test; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.67 to -0.02]
Statistical Analysis 3: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 3; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -1.29, 95% CI 2-sided [-1.68 to -0.91]
Statistical Analysis 4: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 4; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -1.80, 95% CI 2-sided [-2.25 to -1.36]
Statistical Analysis 5: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 5; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.24, 95% CI 2-sided [-2.78 to -1.69]
Statistical Analysis 6: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 6; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.08, 95% CI 2-sided [-2.70 to -1.45]
Statistical Analysis 7: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 7; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.97, 95% CI 2-sided [-3.84 to -2.10]

14. Secondary Outcome: Post Otrivine Use Score for Additional Health Related QoL Factors: Snoring
Description: Health related QoL factors were assessed using questions related to snoring, alertness, self-consciousness about how participants sound, smell, taste, self-consciousness around people, energy, and motivation. Participants rated their response to questions on a scale ranging from 0 to 7, where 0= Not at all and 7= Severely. The minimum and maximum score for each question was 0 and 7 respectively, where lower score indicated improvement.
Time Frame: Days 1, 2, 3, 4, 5, 6, and 7
Population: mITT population. Here, overall number analyzed is defined as the number of participants with data available for analysis for this outcome measure. Only those participants with data available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride)
Number analyzed (Participants) | 73
score on a scale
  Day 1 | 2.8 (2.11)
  Day 2: number analyzed (Participants) | 71
  Day 2 | 2.4 (2.04)
  Day 3: number analyzed (Participants) | 69
  Day 3 | 1.9 (1.95)
  Day 4: number analyzed (Participants) | 61
  Day 4 | 1.4 (1.79)
  Day 5: number analyzed (Participants) | 41
  Day 5 | 1.4 (1.63)
  Day 6: number analyzed (Participants) | 27
  Day 6 | 1.4 (1.58)
  Day 7: number analyzed (Participants) | 25
  Day 7 | 1.2 (1.44)
Statistical Analysis 1: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 1; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -1.88, 95% CI 2-sided [-2.33 to -1.43]
Statistical Analysis 2: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 2; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.45, 95% CI 2-sided [-2.90 to -2.01]
Statistical Analysis 3: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 3; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.90, 95% CI 2-sided [-3.41 to -2.39]
Statistical Analysis 4: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 4; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -3.30, 95% CI 2-sided [-3.82 to -2.77]
Statistical Analysis 5: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 5; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.95, 95% CI 2-sided [-3.53 to -2.37]
Statistical Analysis 6: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 6; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -3.26, 95% CI 2-sided [-3.98 to -2.53]
Statistical Analysis 7: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 7; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -3.12, 95% CI 2-sided [-4.08 to -2.16]

15. Secondary Outcome: Post Otrivine Use Score for Additional Health Related QoL Factors: Alertness
Description: as for outcome 14
Time Frame: Days 1, 2, 3, 4, 5, 6, and 7
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride)
Number analyzed (Participants) | 98
score on a scale
  Day 1 | 2.1 (1.94)
  Day 2: number analyzed (Participants) | 97
  Day 2 | 1.8 (1.81)
  Day 3: number analyzed (Participants) | 92
  Day 3 | 1.6 (1.80)
  Day 4: number analyzed (Participants) | 82
  Day 4 | 1.1 (1.61)
  Day 5: number analyzed (Participants) | 59
  Day 5 | 0.8 (1.17)
  Day 6: number analyzed (Participants) | 39
  Day 6 | 0.8 (1.14)
  Day 7: number analyzed (Participants) | 30
  Day 7 | 0.8 (1.18)
Statistical Analysis 1: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 1; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -1.72, 95% CI 2-sided [-2.14 to -1.31]
Statistical Analysis 2: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 2; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.12, 95% CI 2-sided [-2.55 to -1.70]
Statistical Analysis 3: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 3; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.30, 95% CI 2-sided [-2.71 to -1.90]
Statistical Analysis 4: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 4; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.76, 95% CI 2-sided [-3.23 to -2.29]
Statistical Analysis 5: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 5; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.85, 95% CI 2-sided [-3.31 to -2.39]
Statistical Analysis 6: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 6; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -3.18, 95% CI 2-sided [-3.72 to -2.64]
Statistical Analysis 7: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 7; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -3.17, 95% CI 2-sided [-3.90 to -2.43]

16. Secondary Outcome: Post Otrivine Use Score for Additional Health Related QoL Factors: Self-conscious About Sound
Description: as for outcome 14
Time Frame: Days 1, 2, 3, 4, 5, 6, and 7
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride)
Number analyzed (Participants) | 98
score on a scale
  Day 1 | 2.2 (1.85)
  Day 2: number analyzed (Participants) | 97
  Day 2 | 2.0 (1.99)
  Day 3: number analyzed (Participants) | 92
  Day 3 | 1.6 (1.76)
  Day 4: number analyzed (Participants) | 82
  Day 4 | 1.4 (1.75)
  Day 5: number analyzed (Participants) | 59
  Day 5 | 1.1 (1.56)
  Day 6: number analyzed (Participants) | 39
  Day 6 | 1.3 (1.69)
  Day 7: number analyzed (Participants) | 30
  Day 7 | 0.9 (1.28)
Statistical Analysis 1: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 1; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -1.98, 95% CI 2-sided [-2.39 to -1.57]
Statistical Analysis 2: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 2; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.24, 95% CI 2-sided [-2.66 to -1.81]
Statistical Analysis 3: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 3; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.73, 95% CI 2-sided [-3.14 to -2.32]
Statistical Analysis 4: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 4; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.91, 95% CI 2-sided [-3.40 to -2.43]
Statistical Analysis 5: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 5; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -3.17, 95% CI 2-sided [-3.68 to -2.66]
Statistical Analysis 6: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 6; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -3.28, 95% CI 2-sided [-4.02 to -2.54]
Statistical Analysis 7: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 7; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -3.47, 95% CI 2-sided [-4.24 to -2.70]

17. Secondary Outcome: Post Otrivine Use Score for Additional Health Related QoL Factors: Smell
Description: as for outcome 14
Time Frame: Days 1, 2, 3, 4, 5, 6 and 7
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride)
Number analyzed (Participants) | 98
score on a scale
  Day 1 | 2.8 (1.89)
  Day 2: number analyzed (Participants) | 97
  Day 2 | 2.4 (1.99)
  Day 3: number analyzed (Participants) | 92
  Day 3 | 1.8 (1.81)
  Day 4: number analyzed (Participants) | 82
  Day 4 | 1.5 (1.65)
  Day 5: number analyzed (Participants) | 59
  Day 5 | 1.2 (1.59)
  Day 6: number analyzed (Participants) | 39
  Day 6 | 1.5 (1.80)
  Day 7: number analyzed (Participants) | 30
  Day 7 | 1.3 (1.70)
Statistical Analysis 1: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 1; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -1.96, 95% CI 2-sided [-2.37 to -1.55]
Statistical Analysis 2: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 2; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.42, 95% CI 2-sided [-2.83 to -2.01]
Statistical Analysis 3: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 3; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.97, 95% CI 2-sided [-3.41 to -2.53]
Statistical Analysis 4: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 4; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -3.34, 95% CI 2-sided [-3.81 to -2.87]
Statistical Analysis 5: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 5; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -3.36, 95% CI 2-sided [-3.84 to -2.87]
Statistical Analysis 6: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Change from Baseline at Day 6; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -3.23, 95% CI 2-sided [-3.91 to -2.56]
Statistical Analysis 7: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 7; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -3.70, 95% CI 2-sided [-4.48 to -2.92]

18. Secondary Outcome: Post Otrivine Use Score for Additional Health Related QoL Factors: Taste
Description: as for outcome 14
Time Frame: Days 1, 2, 3, 4, 5, 6 and 7
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride)
Number analyzed (Participants) | 98
score on a scale
  Day 1 | 2.4 (2.01)
  Day 2: number analyzed (Participants) | 97
  Day 2 | 2.1 (2.03)
  Day 3: number analyzed (Participants) | 92
  Day 3 | 1.8 (1.91)
  Day 4: number analyzed (Participants) | 82
  Day 4 | 1.4 (1.67)
  Day 5: number analyzed (Participants) | 59
  Day 5 | 1.3 (1.65)
  Day 6: number analyzed (Participants) | 39
  Day 6 | 1.3 (1.78)
  Day 7: number analyzed (Participants) | 30
  Day 7 | 1.3 (1.67)
Statistical Analysis 1: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 1; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -1.76, 95% CI 2-sided [-2.17 to -1.34]
Statistical Analysis 2: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 2; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.09, 95% CI 2-sided [-2.51 to -1.67]
Statistical Analysis 3: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 3; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.41, 95% CI 2-sided [-2.86 to -1.97]
Statistical Analysis 4: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 4; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.74, 95% CI 2-sided [-3.22 to -2.27]
Statistical Analysis 5: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 5; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.73, 95% CI 2-sided [-3.30 to -2.16]
Statistical Analysis 6: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 6; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.87, 95% CI 2-sided [-3.56 to -2.19]
Statistical Analysis 7: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 7; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -3.20, 95% CI 2-sided [-4.01 to -2.39]

19. Secondary Outcome: Post Otrivine Use Score for Additional Health Related QoL Factors: Self-conscious Around People
Description: as for outcome 14
Time Frame: Day 1, 2, 3, 4, 5, 6 and 7
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride)
Number analyzed (Participants) | 98
score on a scale
  Day 1 | 2.3 (1.96)
  Day 2: number analyzed (Participants) | 97
  Day 2 | 1.7 (1.76)
  Day 3: number analyzed (Participants) | 92
  Day 3 | 1.6 (1.70)
  Day 4: number analyzed (Participants) | 82
  Day 4 | 1.1 (1.61)
  Day 5: number analyzed (Participants) | 59
  Day 5 | 1.0 (1.40)
  Day 6: number analyzed (Participants) | 39
  Day 6 | 1.0 (1.50)
  Day 7: number analyzed (Participants) | 30
  Day 7 | 0.8 (1.37)
Statistical Analysis 1: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 1; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -1.93, 95% CI 2-sided [-2.35 to -1.51]
Statistical Analysis 2: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 2; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.60, 95% CI 2-sided [-3.00 to -2.20]
Statistical Analysis 3: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 3; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.65, 95% CI 2-sided [-3.09 to -2.22]
Statistical Analysis 4: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 4; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -3.07, 95% CI 2-sided [-3.53 to -2.62]
Statistical Analysis 5: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 5; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -3.25, 95% CI 2-sided [-3.76 to -2.75]
Statistical Analysis 6: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 6; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -3.41, 95% CI 2-sided [-4.04 to -2.78]
Statistical Analysis 7: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 7; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -3.47, 95% CI 2-sided [-4.30 to -2.64]

20. Secondary Outcome: Post Otrivine Use Score for Additional Health Related QoL Factors: Energy
Description: as for outcome 14
Time Frame: Days 1, 2, 3, 4, 5, 6 and 7
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride)
Number analyzed (Participants) | 98
score on a scale
  Day 1 | 3.1 (2.02)
  Day 2: number analyzed (Participants) | 97
  Day 2 | 2.5 (2.06)
  Day 3: number analyzed (Participants) | 92
  Day 3 | 2.1 (1.87)
  Day 4: number analyzed (Participants) | 82
  Day 4 | 1.8 (1.94)
  Day 5: number analyzed (Participants) | 59
  Day 5 | 1.4 (1.54)
  Day 6: number analyzed (Participants) | 39
  Day 6 | 1.2 (1.44)
  Day 7: number analyzed (Participants) | 30
  Day 7 | 1.0 (1.30)
Statistical Analysis 1: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 1; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.07, 95% CI 2-sided [-2.49 to -1.66]
Statistical Analysis 2: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 2; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.76, 95% CI 2-sided [-3.20 to -2.33]
Statistical Analysis 3: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 3; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -3.21, 95% CI 2-sided [-3.63 to -2.78]
Statistical Analysis 4: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 4; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -3.49, 95% CI 2-sided [-3.98 to -3.00]
Statistical Analysis 5: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 5; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -3.83, 95% CI 2-sided [-4.33 to -3.33]
Statistical Analysis 6: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 6; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -4.05, 95% CI 2-sided [-4.65 to -3.46]
Statistical Analysis 7: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 7; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -4.13, 95% CI 2-sided [-4.81 to -3.46]

21. Secondary Outcome: Post Otrivine Use Score for Additional Health Related QoL Factors: Motivation
Description: as for outcome 14
Time Frame: Days 1, 2, 3, 4, 5, 6 and 7
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride)
Number analyzed (Participants) | 98
score on a scale
  Day 1 | 2.9 (2.19)
  Day 2: number analyzed (Participants) | 97
  Day 2 | 2.4 (1.92)
  Day 3: number analyzed (Participants) | 92
  Day 3 | 2.0 (1.90)
  Day 4: number analyzed (Participants) | 82
  Day 4 | 1.7 (1.89)
  Day 5: number analyzed (Participants) | 59
  Day 5 | 1.4 (1.61)
  Day 6: number analyzed (Participants) | 39
  Day 6 | 1.2 (1.54)
  Day 7: number analyzed (Participants) | 30
  Day 7 | 1.1 (1.49)
Statistical Analysis 1: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 1; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.21, 95% CI 2-sided [-2.66 to -1.77]
Statistical Analysis 2: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 2; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -2.73, 95% CI 2-sided [-3.15 to -2.31]
Statistical Analysis 3: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 3; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -3.16, 95% CI 2-sided [-3.60 to -2.73]
Statistical Analysis 4: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 4; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -3.52, 95% CI 2-sided [-4.00 to -3.05]
Statistical Analysis 5: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 5; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -3.73, 95% CI 2-sided [-4.19 to -3.27]
Statistical Analysis 6: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 6; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -4.00, 95% CI 2-sided [-4.55 to -3.45]
Statistical Analysis 7: Comparison: Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride); Day 7; Test type: Other; p < .0001, Student's paired t-test; Mean Difference (Final Values) = -4.07, 95% CI 2-sided [-4.74 to -3.39]

ADVERSE EVENTS:
Time Frame: From first dose of study product administration up to Day 7
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study product including any washout or lead-in product (or medical device), whether or not considered related to the study product, including any washout or lead-in product (or medical device). All-Cause Mortality included all randomized participants. Serious and Other AEs: Safety population included all participants who used study product at least once.
Arm/Group | Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride)
All-Cause Mortality (participants affected / at risk) | 0/136
Serious Adverse Events (participants affected / at risk) | 0/102
Other Adverse Events (participants affected / at risk) | 6/102
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Otrivine Congestion Relief 0.1% Nasal Spray (Xylometazoline Hydrochloride) (N=102)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1
Eye Pruritus (Eye disorders) | 1
Lacrimation Increased (Eye disorders) | 1
Headache (Nervous system disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Sinusitis (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
HALEON agreements may vary with individual investigators but will not prohibit any investigator from publishing. HALEON supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/48/NCT05556148/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-04): https://cdn.clinicaltrials.gov/large-docs/48/NCT05556148/SAP_001.pdf